CLINICAL TRIAL: NCT00651768
Title: A 52 wk Randomized, Doubleblind, Single Dummy, Parallel Group Multicenter Phase 3 Study Comparing the Long Term Safety of Symbicort pMDI 4x160/4.5mcg Bid to SymbicortpMDI 2x160/4.5mcg Bid & Budesonide HFA pMDI 4x160mcg Bid in Adult and Adolescent Subjects With Asthma
Brief Title: Titratable Dosing in Moderate to Severe Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-039-0728; D5896C00728
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: asthma; adults; adolescents; safety; Symbicort; budesonide/formoterol; budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: budesonide/formoterol
- 2 (Sham Comparator)
  Interventions: Drug: Symbicort pMDI + budesonide HFA pMDI

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: Symbicort pMDI + budesonide HFA pMDI — Symbicort 2 X 160/4.5mcg & budesonide HFA pMDI 4 X 160mcg
  Arms: 2

SUMMARY:
The purpose of this study is to compare the long term safety of Symbicort with budesonide alone, in adolescents and adults with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma and baseline lung function tests, symptoms and medication use as determined by the protocol
* Required and received treatment with inhaled corticosteroids within the timeframe and doses specified in the protocol

Exclusion Criteria:

* Has required treatment with non-inhaled corticosteroids within previous 30 days, has sensitivity to drugs specified in the protocol or requires treatment with a beta-blocker.
* Has had cancer within previous 5 years or has a condition that may put the patient at risk in this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2003-08; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations, ECG and Holter monitors, lung function, adverse events, requirement of other asthma therapies and other routine safety assessments. | 7 assessments within 12 month treatment period

SECONDARY OUTCOMES:
To measure changes in lung function tests, patient reported outcomes and usage of medical resource | 7 assessments within 12 month treatment period
Blood levels of budesonide and formoterol | 10 blood samples taken at 1 visit in a sub-set of patients

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162